CLINICAL TRIAL: NCT05158049
Title: Longitudinal Observation and Assessment of the Suprachoroidal Retinal Prostheses
Brief Title: Longitudinal Study of a Bionic Eye
Status: Enrolling by invitation | Type: Observational
Sponsor: Center for Eye Research Australia (Other)
Collaborators: The Bionics Institute of Australia (Other); Australian National University (Other); Commonwealth Scientific and Industrial Research Organisation, Australia (Other Government); Bionic Vision Technologies (Unknown)
Responsible Party: Sponsor
Other Study IDs: 75829
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Retinitis Pigmentosa; Choroideremia
MeSH Terms: conditions — Retinitis Pigmentosa; Choroideremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a longitudinal observational study with participants who have been implanted with the suprachoroidal retinal prosthesis.

DETAILED DESCRIPTION:
To observe and assess visual, orientation and mobility behavior with primary and adjunct vision processing (AVP) methods that may enhance the performance with the suprachoroidal retinal prosthesis (ScRP). To investigate the effectiveness of primary and AVP methods in the laboratory and real-world environments with the ScRP. Assess structural and functional ScRP stability with objective and subjective assessments. Record participant experiences and feedback with the ScRP.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide signed informed consent;
* Implanted with a suprachoroidal retinal prosthesis;
* Be available for the study visits;
* Willing to comply with study assessments;
* In good general health and mobile.

Exclusion Criteria:

* Medical condition that prohibits mobility;
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who were implanted with a suprachoroidal retinal prosthesis.
Sampling Method: Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2026-12-09 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of vision processing method in the laboratory. | 5 years.
  Measure effectiveness of of the vision processing method via observational and quantitative data.
Effectiveness of vision processing method in the 'real world' featured environment. | 5 years.
  Measure the effectiveness of the vision processing method via observational qualitative and quantitative data in participant 'real world' featured environment.

SECONDARY OUTCOMES:
Device stability and functionality. | 5 years.
  Monitor device stability with routine ophthalmic imaging, impedance and threshold testing.
Participant experience. | 5 years
  Document participant anecdotal experience with the VP method in 'real world' environments.
Participant interview. | 5 years
  Interview participants to capture participant experience with the ScRP, determine differences in functional outcomes and utilise this information to improve assessment of functional outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Penelope J Allen, FRACO, FRACS, Principal Investigator — Center for Eye Research Australia
Locations (1):
- Centre for Eye Research Australia, Melbourne E., Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Moussallem L, Lombardi L, McGuinness MB, Kolic M, Baglin EK, Jin R, Habili N, Kvansakul J, Titchener SA, Abbott CJ, Walker JG, Allen PJ, Petoe MA, Barnes N. Navigational outcomes with a depth-based vision processing algorithm in a second-generation suprachoroidal retinal prosthesis. J Neural Eng. 2025 Apr 24;22(2). doi: 10.1088/1741-2552/adc83a. PMID 40174607
- See also: Study of a Suprachoroidal Retinal Prosthesis — https://clinicaltrials.gov/ct2/show/NCT03406416
- See also: Pilot Study of a Suprachoroidal Retinal Prosthesis — https://clinicaltrials.gov/ct2/show/NCT01603576